CLINICAL TRIAL: NCT01216150
Title: Impact of Combination of Clopidogrel With Aspirin on Postoperative Bleeding and Platelets Functions in Coronary Surgical Patients Treated Prophylactically With Tranexamic Acid: the ICARE Study.
Brief Title: Impact of Combination of Clopidogrel With Aspirin on Postoperative Bleeding in Coronary Surgical Patients
Acronym: ICARE
Status: Completed | Type: Observational
Sponsor: Groupe Hospitalier Pitie-Salpetriere (Other)
Responsible Party: AMOUR julien, Hôpital Pitié Salpêtrière, Paris, France
Other Study IDs: ICARE Study
Record Dates: First submitted 2010-10-06; First posted 2010-10-07 (Estimated); Last update posted 2011-06-23 (Estimated); Status verified 2010-10

CONDITIONS: Coronary Surgery; Hemorrhage
Keywords: antifibrinolytic drug; coronary surgery; hemorrhage; aspirin; clopidogrel
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- aspirin: group treated with aspirin alone
- aspirin clopidogrel: Goup treated with aspirin and clopidogrel

SUMMARY:
Aims Aspirin combined with clopidogrel is the treatment of choice for acute coronary syndromes. Although the maintenance of aspirin until surgery does not affect postoperative bleeding after coronary artery bypass graft (CABG) surgery, the latter may be dramatically increased when clopidogrel is continued over a period of 5 days preoperatively. Methods and results: This prospective observational study will include 136 consecutive patients scheduled for first-time CABG. Postoperative bleeding and blood transfusion requirements will be compared (non inferiority)between patients pretreated during a period of 5 days prior surgery by either aspirin alone or combined with clopidogrel. Tranexamic acid will be systematically used in all these patients considered as high risk for bleeding.

In concusion, this study has to to test the hypothesis that with tranexamic acid also, bleeding in the aspirin + clopidogrel group is not 25% more important than in the aspirin alone group after CABG surgery, according to the previous study using aprotinin.

DETAILED DESCRIPTION:
Impact of combination of clopidogrel with aspirin on postoperative bleeding and platelets functions in coronary surgical patients treated prophylactically with tranexamic acid.

Introduction Major cardiac events are known to be reduced in patients with acute coronary syndrome by an association of aspirin with clopidogrel (1)(2). In cardiac surgery as well, aspirin treatment has been shown to reduce major cardio-vascular events and mortality in postoperative period after coronary artery bypass grafting (CABG) without any increase of postoperative bleeding (3)(4). In a recent study performed in our department, Ouattara and al. have shown in cardiac surgery that the combination of aspirin with clopidogrel does not increase postoperative bleeding, transfusion or surgical reexploration after CABG when aprotinin is used during surgery, by comparison to aspirin alone (5). In conclusion, the authors suggested no disruption of aspirin and clopidogrel when patients are treated with this association before surgery. Unfortunately, since the trials of Mangano and al. (6) and of the BART investigators (7), aprotinin, a plasmin inhibitor derived from bovine lung tissues, has been withdrawn for safety reasons. Therefore, physicians are restrained to use instead tranexamic acid, a synthetic molecule that inhibits conversion of the inactive plasminogen to plasmin, to minimize bleeding and to reduce exposure to blood products.

The aim of this study is to test the hypothesis that with tranexamic acid also, bleeding in the aspirin + clopidogrel group is not 25% more important than in the aspirin alone group after CABG surgery, according to the previous study using aprotinin. In the present study, the functionality of the platelets tested before the surgical procedure will be compared to level of the first 24 hours bleeding.

Methods Selection of patients This prospective observational study will be conducted at the Institute of Cardiology in the Pitié-Salpêtrière Hospital, Paris, France. It is planned to start in december 2009 to november 2010. Care of patients will conform to standard procedures currently used in our institute, which will not be modified by the study. Platelet function will be measured in residual blood samples, after ethical committee approval (Comité de Protection des Personnes VI - Ile de France). A written informed consent is not resquested from patients. Nevertheless, written information will be delivered for each of them. During the planned 11 months of investigation, all patients undergoing isolated first-time coronary artery by-pass grafting will be enrolled. Patients admitted for emergency procedure, following failed percutaneous transluminal coronary angioplasty and off-pump coronary surgery, will be excluded. Because antithrombotic therapy management may differ during the postoperative period, we will exclude patients in whom a mechanical support or intra-aortic balloon pump will be required for a difficult weaning from cardiopulmonary bypass. Finally, we will exclude all patients who will not have received any oral antiplatelet agents within 5 days prior surgery, those who will have been preoperatively exposed to platelet glycoprotein IIb/IIIa inhibitors, and those with history of haematological disease. Patients treated with aspirin and clopidogrel and in whom clopidogrel will be stopped more than 5 days before surgery will also be excluded.

Intraoperative management Patients will be monitored with arterial and central venous catheterizations. All patients will be considered at high risk for postoperative bleeding as they will receive at least one antiplatelet agent and therefore will be administered tranexamic acid (Exacyl®, Sanofi-Aventis, Paris, France) according to the following standardized protocol: infusion of 10 mg/kg for 20 minutes during anaesthesia induction, followed by a continuous infusion until the end of surgery, according to renal function of patients as described by Nuttall et al. (8) (See table below). The rest of intraoperative management will be the same as previously described by Ouattara and al. (5). Briefly, before aortic cannulation, an initial loading dose of heparin will be directly administered by the surgeon into the right atrium and then anticoagulation will be maintained by additional bolus during the extracorporeal circulation. Non-pulsatile cardiopulmonary bypass will be ensured at a flow of 2.4 L/min/m2. The temperature of systemic perfusion during cardiopulmonary bypass (hypothermia <32°C, mild hypothermia 32-36°C, and normothermia >36°C) will be left to the discretion of the attending surgeon. After discontinuation of the cardiopulmonary bypass, heparin will be neutralized by protamin sulfate (0.008-0.01 mg/IU of total heparin dose intraoperatively used). Intraoperative cell salvage will be systematically used (Electa, Dideco, Mirandola, Italy). The use of inotropes for difficult weaning from cardiopulmonary bypass will be left to the discretion of the attending anaesthesiologist. Discontinuation of the cardiopulmonary bypass will be done when central body temperature (estimated by vesical temperature) will be above 35°C.

Creatinine Tranexamic acid dose < 140 µmol/L 2 mg/kg/h 140 - 290 µmol/L 1,5 mg/kg/h 291 - 580 µmol/L 1 mg/kg/h > 580 µmol/L 0,5 mg/kg/h Table: dosing of tranexamic acid according to renal function, from Nuttall and al. (8)

Postoperative antithrombotic therapy The early postoperative antithrombotic therapy will be based on intravenous bolus of 100 mg aspirin given 6 h after the arrival in intensive care unit, as previously described. The day after surgery, enoxaparin 40 mg will be given once daily subcutaneously. The perioperative blood transfusion will be done according to the French National recommendations (9). In patients preoperatively treated by combined antiplatelet therapy, clopidogrel will be re-introduced the day after the surgery.

Antiplatelet therapy efficiency monitoring

Pre-operative platelet function will include :

1. Platelet aggregation tests Aggregation studies will be performed within 3 hours after blood collection by Pascale Gaussem (INSERM U765, HEGP), as published elsewhere (10). Aggregation tests are performed on platelet-rich plasma adjusted to 250x109/L platelets using the following agonists: arachidonic acid 1.5 and 2 mmol/l (Helena biosciences Europe) to explore aspirin effect, Horm collagen 1 µg/ml to explore global platelet function (Nycomed Pharma) and ADP 10 and 20 µmol/l (Biopool) to explore clopidogrel effect.

   A whole blood platelet impedance aggregation test will be performed using the Multiplate® (IL) device and various agonists.
2. Flow cytometry assays VASP phosphorylation: clopidogrel effect VASP (vasodilator-stimulated phosphoprotein) is measured in whole blood with a commercial kit (Platelet VASP; Diagnostica Stago, Biocytex) on a FACScan flow cytometer (Becton Dickinson). The results are expressed as the platelet reactivity index (PRI, %).

Secretory capacity of platelets Platelet secretion will be tested by their capacity to expose surface P-selectin (CD62P) after activation with the thrombin receptor peptide agonist (TRAP) as published elsewhere.

Circulating platelet-leukocyte complexes Circulating activated platelets form complexes with leukocytes via CD62P-PSGL interaction. These complexes are quantified on a population of 5000 leukocytes. Complexes are identified by flow cytometry as the cell population stained with both anti-CD41-PE (platelet marker) and anti-CD45-FITC (leukocyte marker) and are expressed as a percentage of total leukocytes.

Endpoints The primary outcome will be the chest blood output during the first 24 hours. Size sample calculation : bleeding with aspirin alone is estimated around 400±200 mL after CABG (5). Excessive bleeding will be defined by an increment of at least 25% of this basal value collected through chest tubes during the first 24 postoperative hours. Secondary outcomes will be the rate of re-exploration for excessive bleeding, transfusion requirement, prolonged mechanical ventilation (>10 h), and intensive care unit length of stay (>72 h).

Statistical analysis With an estimated distribution of 60% / 40% between aspirin alone and aspirin + clopidogrel groups and assuming an alpha risk of 0.05 and a beta risk of 0.20 and a mean amount of postoperative bleeding after CABG in the aspirin-alone group of 400 +/- 200 mL, we calculate that at least 136 patients at all (85 in aspirin alone and 51 in aspirin + clopidogrel) are required to demonstrate that the amount of bleeding in the aspirin+clopidogrel was not more than 25% increased compared to the bleeding in aspirin alone group (non inferiority study).

Lastly, supposing a few patients lost to follow up and several technical problems after sample collection in platelets function analysis, the final number of patients to include is estimated to be 150 and thus the predicted duration of inclusion will be 44 weeks.

Categorical variables will be compared using Fisher's exact test and continuous variables using the Mann-Witney U test. The postoperative hemoglobin levels and platelet counts will be compared using analysis of variance for repeated measurements completed using a Newman-Keuls test for post-test analysis.

Since this study is not randomized, the patients receiving clopidogrel preoperatively may not have the same peri-operative risk of excessive bleeding than those who do not. Therefore, we will perform separate multivariable risk adjustment to analyze the perioperative risk associated with clopidogrel treatment. For each patient, a propensity score, indicating the likelihood of having clopidogrel, will be calculated. The propensity score-matched analysis will allows us to determine whether preoperative clopidogrel therapy is independently associated with an increased risk of excessive postoperative bleeding. All preoperative variables as well as second-order interaction terms will be entered into the model. Calibration and discrimination of the final logistic model will be assessed using the Hosmer-Lemeshow statistics and the receiver operating characteristic curve, respectively. Comparison of mean bleeding between several groups (according to propensity score quintiles) will be performed using analysis of variance.

Data will be expressed as mean+SD, median, and 5th-95th percentiles or percentage of patients as specified. All P-values will be two tailed and a value less than 0.05 will be required to reject the null hypothesis.

References

1. Fox KAA, Mehta SR, Peters R, Zhao F, Lakkis N, Gersh BJ, Yusuf S. Benefits and risks of the combination of clopidogrel and aspirin in patients undergoing surgical revascularization for non-ST-elevation acute oronary syndrome. The clopidogrel in unstable angina to prevent recurrent ischaemic events (CURE) trial. Circulation. 2004, Vol. 110, pp. 1202-1208.
2. The clopidogrel in unstable angina to prevent recurrent ischaemic events trials investigators. Effects of clopidogrel in addition to aspirin in patients with acute coronary syndromes without ST-segment elevation. N Engl J Med. 2001, 345, pp. 494-502.
3. Tuman KJ, McCarthy RJ, O'Connor CJ, McCarthy WE, Ivankovich AD. Aspirin does not increase allogenic blood transfusion in reoperative coronary artery surgery. Anesth Analg. 1996, Vol. 83, pp. 1178-1184.
4. Dacey LJ, Munoz JJ, Johnson ER, Leavitt BJ, Maloney CT, Morton JR,Olmstead EM, Birkmeyer JD, O'Connor GT for the Northern New England Cardiovascular. Effect of preoperative aspirin use on mortality in coronary artery bypass grafting patients. Ann Thorac Surg. 2000, Vol. 70, pp. 1986-1990.
5. Ouattara A, Bouzguenda H, Le Manach Y, Léger Ph, Mercadier A, Leprince P, Bonnet N, Montalescot G, Riou B, Coriat P. Impact of aspirin with or without clopidogrel on postoperative bleeding and blood transfusion in coronary surgical patients treated prophylactically with a low-dose of aprotinin. Eur Heart J. 2007, Vol. 28, pp. 1025-1032.
6. Mangano DT, Tudor IC, Dietzel C, Group, Multicenter Study of Preoperative Ischemia Research et Fondation, Ischemia Research and Education. The risk associated with aprotinin in cardiac surgery. N Engl J Med. 2006, Vol. 354(4), pp. 353-65.
7. Fergusson DA, Hébert PC, Mazer CD, Fremes S, MacAdams C, Murkin JM, Teoh K, Duke PC, Arellano R, Blajchman MA, Bussières JS, Côté D, Karski J, Martineau R, Robblee JA, Rodger M, Welles G, Clinch J, Pretorius R, for the BART investigator. A comparison of aprotinin and lysine analogues in high risk cardiac surgery. N Engl J Med. 2008, Vol. 358, 22, pp. 2319-2331.
8. Nuttal GAl, Gutierrez MC, Dewey JD. A Preliminary Study of a New Tranexamic Acid Dosing Schedule for Cardiac Surgery. Journal of Cardiothoracic and Vascular Anesthesia. 2008, Vol. 22, 2, pp. 230-235.
9. Agence Française de Sécuité Sanitaire des Produits de Santé (AFSSAPS). Transfusion of erythrocytes substitutes: products, indications, alternatives. General methods and recommendations. Transfus Clin Biol. 2002, Vol. 9, pp. 333-356.
10. Dupont A, Fontana P, Bachelot-Loza C, Reny JL, Bieche I, Desvard F, et al. An intronic polymorphism in the PAR-1 gene is associated with platelet receptor density and the response to SFLLRN. Blood 2003;101:1833-40.

ELIGIBILITY:
Inclusion Criteria:

* all patients undergoing isolated first-time coronary artery by-pass grafting will be enrolled.

Exclusion Criteria:

* patient who do not want to be include
* pregnant
* patient < 18 yrs old
* emergency procedure with failed percutaneous transluminal coronary angioplasty
* off-pump coronary surgery
* patients in whom a mechanical support (ECMO) or intra-aortic balloon pump will be required for a difficult weaning from cardiopulmonary bypass
* patients who will not have received any oral antiplatelet agents within 5 days prior surgery
* patient who will be preoperatively exposed to platelet glycoprotein IIb/IIIa inhibitors
* Patients treated with aspirin and clopidogrel and in whom clopidogrel will be stopped more than 5 days before surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: During the planned 11 months of investigation, all patients undergoing isolated first-time coronary artery by-pass grafting will be enrolled. Patients admitted for emergency procedure, following failed percutaneous transluminal coronary angioplasty and off-pump coronary surgery, will be excluded. Because antithrombotic therapy management may differ during the postoperative period, we will exclude patients in whom a mechanical support or intra-aortic balloon pump will be required for a difficult weaning from cardiopulmonary bypass. Finally, we will exclude all patients who will not have received any oral antiplatelet agents within 5 days prior surgery, those who will have been preoperatively exposed to platelet glycoprotein IIb/IIIa inhibitors, and those with history of haematological disease. Patients treated with aspirin and clopidogrel and in whom clopidogrel will be stopped more than 5 days before surgery will also be excluded.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2009-12; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
chest blood output during the first 24 hours | 24 hours postoperative
  Chest blood collected through chest tubes during the first 24 postoperative hours.

SECONDARY OUTCOMES:
the rate of re-exploration for excessive bleeding, transfusion requirement, prolonged mechanical ventilation (>10 h), and intensive care unit length of stay (>72 h). | During critical care unit hospitalisation

CONTACTS AND LOCATIONS:
Overall Officials: Julien Amour, MD.PhD, Study Director — Groupe Hospitalier Pitie-Salpetriere
Locations (1):
- Hopital Pitié Salpêtrière, Paris, France